CLINICAL TRIAL: NCT04825132
Title: Aged European Population QUality of Life in Infectious Diseases
Brief Title: Infectious Diseases in Aged Population
Acronym: AEQUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC20.248
Record Dates: First submitted 2021-02-09; First posted 2021-04-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Infections in Old Age; Bacteremia
Keywords: functional dependency; quality of life; elderly people; respiratory infection; bacteraemia; disability
MeSH Terms: conditions — Bacteremia; Respiratory Tract Infections; Toxemia

STUDY DESIGN:
Intervention Model Description: Longitudinal case-control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacteremia and/or acute respiratory infection (Experimental): Hospitalized in a study center (emergency department, infectious disease, internal medicine or geriatric hospital wards…) for with bacteraemia and/or acute respiratory infection
  Interventions: Other: Geriatric assessment tools
- Without suspicion of infection (Active Comparator): The control patient will undergo the exact same procedures as the case patient described before except for the blood and respiratory sample part. • The typical control patient will be of the same age (+/- 3 years, but aged above 65 years), same sex, without suspicion of infection and hospitalized during the past or upcoming month in the same centre. There will be 2 controls for one case.
  Interventions: Other: Geriatric assessment tools

INTERVENTIONS:
Other: Geriatric assessment tools — Multidimensional Prognostic Index (Living status, medications, ADL, IADL, MMSE mental evaluation, ESS pressure sores, chronic disease, nutritional assessment)

SUMMARY:
The increasing number of persons >65 years of age form a special population at risk for nosocomial and other health care-associated infections. The vulnerability of this age group is related to impaired host defenses such as diminished cell-mediated immunity. Lifestyle considerations, e.g., travel and living arrangements, and residence in nursing homes, can further complicate the clinical picture. The magnitude and diversity of health care-associated infections in the aging population are generating new arenas for prevention and control efforts.

Common infections leading to hospitalizations in this age group result in respiratory infections and bacteraemia and the impact of these infections on the quality of life and disability in aged populations has not been accurately quantified in a European setting.

This study aims to capture and quantify the impact of infectious diseases on quality of life in an aged population.

DETAILED DESCRIPTION:
An emerging public health challenge is to protect the growing ageing population from infectious diseases, which can significantly impact the quality of life of those affected.

The vulnerability of this age group is related to impaired host defenses such as diminished cell-mediated immunity. Lifestyle considerations, e.g., travel and living arrangements, and residence in nursing homes, can further complicate the clinical picture.

The increasing number of persons >65 years of age form a special population at risk for nosocomial and other health care-associated infections. The vulnerability of this age group is related to impaired host defenses such as diminished cell-mediated immunity. Lifestyle considerations, e.g., travel and living arrangements, and residence in nursing homes, can further complicate the clinical picture. The magnitude and diversity of health care-associated infections in the aging population are generating new arenas for prevention and control efforts.

Common infections leading to hospitalizations in this age group result in respiratory infections and bacteraemia and the impact of these infections on the quality of life in aged populations has not been accurately quantified in a European setting.

This study aims to capture and quantify the impact of infectious diseases on quality of life in an aged population.

The IMI European public-private partnership created the VITAL project (Vaccines and infectious diseases in the Ageing populations) to assess the infectious diseases burden and mechanisms of immunosenescence in the ageing populations. This aims to provide evidence-based knowledge on vaccination strategies to establish healthy ageing. The project articulates around five work packages and this study comes within the frame of the first one. The expected results of this work combine with and complete the retrospective assessment already done on the available datasets/databases.

The decreased efficiency of the cell-mediated immunity and more generally the immunosenescence make the ageing population prone to harming infectious diseases. That combined with the growth of the ageing populations make healthy ageing a major and current challenge to address. The common infections leading to hospitalizations in this age groups include respiratory infections and bacteremia.

Acute respiratory infections (ARI) are a leading cause of hospitalizations and death in the aged adult population. They can be caused by viruses (Influenza for instance), bacteria (Streptococcus pneumoniae for instance) and fungi, with either a single or a co-infection. Viruses and bacteria have a comparable share in causing ARI, and a significant part of them are vaccine preventable pathogens. Although the burden of ARI is highest in the ageing population, vaccine effectiveness is the lowest in this vulnerable population, mostly because of immunosenescence. This issue can be tackled by increasing vaccine coverage and efficiency and developing vaccines and treatments for the pathogens leaving physicians with limited prevention and therapeutic options.

Bacteremia is defined by the presence of viable bacteria in the circulating blood generally causing fever, chills, tachycardia, tachypnea, and sometimes requiring hospitalization. It increases morbidity and has a high mortality rate in all ageing populations. It is mostly caused by Gram negative (E. Coli, Proteus mirabilis, Klebsiella) but also by Gram positive bacteria (Staphylococcus aureus). Along with its high burden in this population, bacteremia is difficult to tackle because of an odd and nonspecific clinical presentation. In addition, bacteremia is associated with comorbidities, underlying diseases and long-term care centres stays. The increasing proportion of antimicrobial resistance such as methicillin-resistant Staphylococcus aureus (MRSA), vancomycin-resistant Staphylococcus aureus (VRSA) or extended spectrum beta-lactamase (ESBL) make complete eradication harder in a given patient and may alter his quality of life in a durable way.

There is a high ARI and bacteremia burden in the aged population in terms of morbidity and mortality. This burden is also believed to be expressed in terms of lower quality of life, and increased frailty and disability and has begun to be assessed in either of the two pathologies.

The impact of ARI and/or bacteremia on those components needs to be assessed in the most comprehensive way as the investigator are facing a specific population: a significant part of the ageing population is already relatively frail. Frailty has been demonstrated as a predictor of bad recovery after an ARI hospitalization in older adults, of being an adverse outcome of acute illness and of being associated with diminished vaccine effectiveness.

The impact of ARI and bacteremia hospitalization on quality of life, frailty and disability in that ageing population has not been assessed in a wide European setting to our knowledge. Filling this data gap will strengthen the evidence-based and guide public health policies concerning vaccination strategies to promote healthy ageing.

ELIGIBILITY:
Inclusion Criteria For Case:

* Hospitalized adults 65 years or older,
* Presenting with bacteremia with positive blood culture (excluding catheter related infections) and/or
* WHO Severe Acute Respiratory Infection (SARI) case definition
* Upper respiratory infection = SARI (fever or history of fever >38°C, cough, onset of the disease within the last 10 days and requires hospitalisation)
* Lower respiratory infection = SARI with confirmed CT/CHR
* Informed consent form signed
* Patient affiliated to social security insurance

Exclusion Criteria For Case:

* Bedridden or terminally ill patient (based upon a threshold of ADL: ≤2 TBD, or CLINICAL FRAILTY SCALE: ≥8 )
* Patients that refuse the 3- and 6-months follow-up phone call assessments
* Patients that will not be able to answer the 3- and 6-months follow-up phone call assessments via a nurse
* Subject in exclusion period for another study,
* Subject who cannot be contacted in an emergency
* Persons referred to in Articles L1121-5 to L1121-8 of the French code of public health (this corresponds to all persons protected: pregnant or parturient women, breastfeeding mothers, persons deprived of liberty by judicial or administrative decision, persons subject to a legal protection measure).

Inclusion Criteria For Controls

* Same age (+/- 3 years)
* same sex,
* without suspicion of infection
* Hospitalized during the past or upcoming month in the same centre.
* Informed consent form signed
* Patient affiliated to social security insurance

Exclusion Criteria For Controls

* Bedridden or terminally ill patient (based upon a threshold of ADL: ≤2 TBD, or CLINICAL FRAILTY SCALE: ≥8 )
* Patients that refuse the 3- and 6-months follow-up phone call assessments
* Patients that will not be able to answer the 3- and 6-months follow-up phone call assessments via a nurse
* Subject in exclusion period for another study,
* Subject who cannot be contacted in an emergency
* Persons referred to in Articles L1121-5 to L1121-8 of the French code of public health (this corresponds to all persons protected: pregnant or parturient women, breastfeeding mothers, persons deprived of liberty by judicial or administrative decision, persons subject to a legal protection measure)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 521 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Evolution of Functional dependency | Baseline and at 6 months
  Change in activities of daily living (ADL) (Scores ADL : 6/6, 0 to 6, best is 6)

SECONDARY OUTCOMES:
Microbial Epidemiology | At 6 months
  Distribution by portal of entry in bacteremia and distribution by infectious agent in respiratory infection and bacteremia
Functional status depending on the infectious causes. | 15 days Before admission, at admission ( whithin 1st day), Up to 10 days, 3 months and 6 months after discharge
  Evolution of Basic and instrumental daily life activities (ADL/IADL) depending on the infectious causes (Scores ADL : 6/6, 0 to 6, best is 6 - IADL score: 8/8 from 0 To 8 best is 8)
Change in Functional status per country and per health care setting | 15 days Before admission, at admission ( whithin 1st day), Up to 10 days, 3 months and 6 months after discharge
  Measure of the change in the functional status: instrumental daily life activities (ADL/IADL) between hospitalization, discharge, M3 and M6 per country and per health care setting (Scores ADL : 6/6, 0 to 6, best is 6 - IADL score: 8/8 from 0 To 8 best is 8)
Medical complications | acute phase Up to 6 months
  Number of medical complications between discharge and M6
Evolution of Frailty | 15 days Before admission, at admission ( whithin 1st day), Up to 10 days, 3 months and 6 months after discharge
  Evolution of Clinical Frailty Scale (from 1 to 9 - Best level 1 worst Level 9 )
Evolution of quality of life | 15 days Before admission, at admission ( whithin 1st day), Up to 10 days, 3 months and 6 months after discharge
  Evolution of EQ 5D - 3L score ( different conditions 0 to 1)
Evolution of quality of life depending on the infectious causes. | 15 days Before admission, at admission ( whithin 1st day), Up to 10 days, 3 months and 6 months after discharge]
  Evolution Evolution of EQ 5D - 3L score ( different conditions 0 to 1) depending on infectious causes
Evolution of Frailty on depending on the infectious causes. | 15 days Before admission, at admission ( whithin 1st day), Up to 10 days, 3 months and 6 months after discharge
  Evolution of Clinical Frailty Scale (from 1 to 9 - Best level 1 worst Level 9 )
Medical complications | acute phase, Up to 10 days, at 3 months and at 6 months
  Type of medical complications requiring or not hospitalization between discharge and M6
Change frailty per country and per health care setting | 15 days Before admission, at admission ( whithin 1st day), Up to 10 days, 3 months and 6 months after discharge
  Measure of the change frailty ( Clinical frailty scale 0-to 9 the best is 0/9)

CONTACTS AND LOCATIONS:
Locations (22):
- France (7):
  - University Hospital Amiens, Amiens
  - Hospital Chambery, Chambéry
  - Groupe Hospitalier Sud Ile de France, Melun
  - Groupement Hospitalier portes de Provence, Montélimar
  - Centre Hospitalier Intercommunal de Villeneuve St Georges., Paris
  - University Hospital Poitiers, Poitiers
  - CHRU Tours, Tours
- Italy (11):
  - Policlinico Universitario Bari, Bari
  - Unità Operativa Complessa di Geriatria-Camposampiero-ULSS 6, Camposampiero
  - S.O.C. Geriatria-Catanzaro, Catanzaro
  - Ospedale Civile di Dolo- ULSS 3 "Serenissima", Dolo
  - Ente Ospedaliero Galliera, Genova
  - Unità Operativa Complessa di Geriatria-Legnago-ULSS 9, Legnago
  - S.C. Geriatria Monza, Monza
  - Azienda Ospedaliera Universitaria Policlinico di Palermo, Palermo
  - Istituto di Geriatria e Gerontologia-Azienda Ospedaliera di Perugia, Perugia
  - UOC Geriatria di Rovigo, Rovigo
  - Malattie infettive - Sanremo, Sanremo
- Spain (4):
  - FCRB - Fundació Clínic per a la Recerca Biomèdica, Barcelona
  - FIBio-HCSC - Fundación para la Investigación Biomédica del Hospital Clínico San Carlos, Madrid
  - FIBio-HRYC - Fundación para la Investigación Biomédica del Hospital Universitario Ramón y Cajal, Madrid
  - Instituto Murciano de Investigación Biosanitaria Virgen de la Arrixaca, Murcia

REFERENCES:
- [Result] Veronese N, Polidori MC, Maggi S, Zamora J, Ruiz-Calvo G, Bangert M, Bourron P, Bausch A, Aviles-Hernandez JD, Lopez-Soto A, Padronguillen D, Lanoix JP, Cruz-Jentoft AJ, Gavazzi G; AEQUI study group. Measuring the impact of hospitalization for infectious diseases on the quality of life of older patients in four European countries: the AEQUI longitudinal matched cohort study (2020-2023). Clin Microbiol Infect. 2025 May;31(5):847-854. doi: 10.1016/j.cmi.2025.01.009. Epub 2025 Jan 20. PMID 39842547